CLINICAL TRIAL: NCT05196542
Title: Abdominal Sacro-hysteropexy Using Proline Mesh Versus Mersilene Tape in Apical Prolapse: a Randomized Controlled Study
Brief Title: Sacro-hysteropexy Using Proline Mesh Versus Mersilene Tape in Apical Prolapse
Acronym: hystropexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Elsibai Anter (Other)
Responsible Party: Sponsor-Investigator, Mohamed Elsibai Anter, principal investigator, Menoufia University
Organization: Menoufia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Simple Mail Transfer Protocol
Record Dates: First submitted 2021-11-26; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Apical Prolapse
Keywords: hystropexy; mesh; mersilene tape

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants will be aware of procedure but unaware of the material used for repair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mersilene tape arm (ETHICON, polyester 5mm double needle) (Experimental): Group 1: patients with apical prolapse who will do Sacro hysteropexy using mersilene tape (polyester 5mm tape with double needle)
  Interventions: Procedure: patients with apical prolapse who will do Sacro hysteropexy using mersilene tape
- polyproline mesh arm (ETHICON, polyprolene mesh) (Other): Group 2: patients with apical prolapse who will do Sacro hysteropexy using poly-proline mesh
  Interventions: Procedure: patients with apical prolapse who will do Sacro hysteropexy using mersilene tape

INTERVENTIONS:
Procedure: patients with apical prolapse who will do Sacro hysteropexy using mersilene tape — comparison between standard poly prolene mesh and the poly ester mersilene tape in Sacro hysteropexy surgical procedure

SUMMARY:
Sacro-hysteropexy Using Proline Mesh Versus Mersilene Tape in Apical Prolapse: a Randomized Controlled Study .Aim of This Study is to Compare Between Using Poly-proline Mesh Versus Mersilene Tape in Abdominal Sacrohysteropexy Repairing Apical Prolapse Stage 2 or More. Outcome Measures: Short Term: investigators Will Evaluate Operative Time, Blood Loss, Hospital Stay Duration, Occurrence of Major Complications, Episodes of Constipation, Urinary Retention and Urinary Tract Infection. Long Term (After 1 year): investigators Will Evaluate Occurrence of Relapse as Well as Late Complications. Local Symptoms, Quality of Life and Sexual Function Will be Evaluated by a Questioner Before and After Surgery

DETAILED DESCRIPTION:
Aim of this study is to compare between using poly-proline mesh versus mersilene tape in abdominal sacrohysteropexy repairing apical prolapse stage ӀӀ or more.

Study Design: This will be a prospective randomized controlled non blind study will include cases with apical prolapse stage 2 or more undergoing abdominal sling between October 2019 and September 2020 in Obstetrics and Gynecology Department, Ain Shams University Hospital and menofia university hospital.

Inclusion Criteria: Women planning sacrohysteropexy for stage 2, 3, or 4 prolapse with or without stress urinary incontinence, Age between 25 and 45, Patient has no uterine pathology necessitate hysterectomy and patient wish to retain her uterus.

Exclusion Criteria:Unfitness for anesthesia, Present pelvic inflammatory disease, Previously identified or suspected massive adhesions between sigmoid and pre-sacral peritoneum, Previous pelvic operations or trial of sling operation.

Prolapse is staged with the use of the pelvic-organ-prolapse quantification (POP-Q) system, a standardized quantitative method for assessment of prolapse. PISQ-12 assesses the sexual function of the woman with prolapse. Urinary incontinence is ruled out by history, examination and urodynamic study.

Randomization using a list of computer-generated random sample into two groups. Group1:patients with apical prolapse who will do Sacro hysteropexy using poly-proline mesh, Group 2:patients with apical prolapse who will do Sacro hysteropexy using mersilene tape.

Technique of procedure: Participants will receive bowel preparation the day before surgery, Prophylactic antibiotics will be given preoperatively.

Abdominal Sacro colpopexy will be performed by laparotomy under general or spinal anesthesia, preferably using a pfannenstiel incision. In group (1) using poly-proline mesh to be fixed to the cervix at the level of the internal os at the uterosacral ligament and the other end to the longitudinal vertebral ligament by non-absorbable sutures. Excess mesh is trimmed and removed.

In group (2) using mersilene tape with double needle to anchor the cervix at the level of the internal os by stitches and then fixed to the longitudinal vertebral ligament. Mesh or tape should be completely covered by peritoneum.

If the patient complains of stress urinary incontinence, it will be managed by trans-obturator tape (TOT) and procedure will be recorded.

Outcome measures: Short term, investigators will evaluate operative time, blood loss, hospital stay duration, occurrence of major complications, episodes of constipation, urinary retention and urinary tract infection.

Long term (after 1year), investigators will evaluate occurrence of relapse as well as late complications. Also local symptoms, quality of life and sexual function will be evaluated by a questioner before and after surgery.

Sample size: Study will include cases with apical prolapse stage ӀӀ or more undergoing abdominal sling between October 2019 and September 2020 in Obstetrics and Gynecology Department, Ain Shams University Hospital and menofia university hospital. On prevalence of 7% and power of 80, number of cases will be estimated of 50 cases in each group.

ELIGIBILITY:
Inclusion Criteria:

* Women planning sacrohysteropexy for stage 2, 3, or 4 prolapse with or without stress urinary incontinence.

  * Age between 25 and 45
  * Patient has no uterine pathology necessitate hysterectomy and patient wish to retain her uterus.

Exclusion Criteria:

Unfitness for anesthesia

* Present pelvic inflammatory disease
* Previously identified or suspected massive adhesions between sigmoid and pre-sacral peritoneum.
* Previous pelvic operations or trial of sling operation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
operative time | 60 minutes
  time taken from start of operation till its end
blood loss | during surgery time
  amount in CC
occurrence of major complications as vascular injury or ureteric injury | during surgery
  injury
urinary retention | 24 hours
  inability to pass urine after catheter removal
hospital stay duration | 24 hours
  how many hours patient stay in hospital after procedure till discharge

SECONDARY OUTCOMES:
occurrence of relapse | 1year after procedure
  recurrence of prolapse
erosion | 1 year after procedure
  exposure of mesh or tape used

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol